CLINICAL TRIAL: NCT05712941
Title: A Multiregional, Randomized, Double-Blinded, Placebo-Controlled Phase 3 Study of Lerociclib With Letrozole, Versus Placebo in Combination With Letrozole, in Participants With Advanced/Metastatic or Recurrent, Grade 1 or Grade 2 Endometrioid Endometrial Carcinoma
Brief Title: Comparison of Letrozole With Lerociclib Versus Letrozole With Placebo Control in Patients With Advanced/Metastatic or Recurrent, Grade 1 or Grade 2 Endometrial Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study is being closed based on corporate changes at EQRx and is not related to any efficacy or safety issues with lerociclib.
Sponsor: EQRx International, Inc. (Industry)
Collaborators: GOG Foundation (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: EQ132-303; GOG-3075 (Other: GOG Foundation); ENGOT-EN17 (Other: European Network of Gynaecological Oncological Trial Groups (ENGOT))
Record Dates: First submitted 2022-10-31; First posted 2023-02-06 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Letrozole 2.5mg by mouth once a day (QD) + Lerociclib 150mg by mouth twice a day (BID) (Experimental)
  Interventions: Drug: Lerociclib; Drug: Letrozole 2.5mg
- Letrozole 2.5mg by mouth once a day (QD) + Placebo (Placebo Comparator)
  Interventions: Drug: Letrozole 2.5mg; Drug: Placebo

INTERVENTIONS:
Drug: Lerociclib — All participants should be treated according to the best-current-practice guidelines and standard of care within each institution or country where the study is conducted.
  Participants will be randomized to receive either lerociclib (administered at 150 mg twice a day (BID) in combination with letrozole (administered at 2.5 mg once a day (QD), or placebo administered in combination with letrozole (2.5 mg QD).
  Participants will also be stratified, using interactive response technology (IRT), by the following randomization strata:
  * Endometrial Cancer (EC) tumor staging (Federation Internationale de Gynecologie et d'Obstetrique [FIGO] Stage III versus FIGO Stage IV versus recurrent)
  * EC tumor grade (Grade 1 versus Grade 2)
  * Geographic location (US versus Europe versus Rest of World)
  Arms: Letrozole 2.5mg by mouth once a day (QD) + Lerociclib 150mg by mouth twice a day (BID)
Drug: Letrozole 2.5mg — All participants should be treated according to the best-current-practice guidelines and standard of care within each institution or country where the study is conducted.
  Participants will be randomized to receive either lerociclib (administered at 150 mg twice daily (BID) in combination with letrozole (administered at 2.5 mg once a day (QD), or placebo administered in combination with letrozole (2.5 mg QD).
  Participants will also be stratified, using interactive response technology (IRT), by the following randomization strata:
  * Endometrial Cancer (EC) tumor staging (Federation Internationale de Gynecologie et d'Obstetrique [FIGO] Stage III versus FIGO Stage IV versus recurrent)
  * EC tumor grade (Grade 1 versus Grade 2)
  * Geographic location (US versus Europe versus Rest of World)
Drug: Placebo — All participants should be treated according to the best-current-practice guidelines and standard of care within each institution or country where the study is conducted.
  Participants will be randomized to receive either lerociclib (administered at 150 mg twice day (BID) in combination with letrozole (administered at 2.5 mg once a day (QD), or placebo administered in combination with letrozole (2.5 mg QD).
  Participants will also be stratified, using interactive response technology (IRT), by the following randomization strata:
  * Endometrial Cancer (EC) tumor staging (Federation Internationale de Gynecologie et d'Obstetrique [FIGO] Stage III versus FIGO Stage IV versus recurrent)
  * EC tumor grade (Grade 1 versus Grade 2)
  * Geographic location (US versus Europe versus Rest of World)
  Arms: Letrozole 2.5mg by mouth once a day (QD) + Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled Phase 3 clinical trial to compare the combination of lerociclib (administered at 150 mg twice a day (BID) with letrozole (administered at 2.5 mg once a day (QD) to that of placebo with letrozole (2.5 mg QD) in female participants with Grade 1 or Grade 2 (ie, low-grade histology) endometrioid endometrial cancer (EC) and advanced/metastatic or recurrent disease.

The study population will consist of female participants with endometrioid EC who are treatment-naïve in the advanced/metastatic setting (ie, the first-line [1L] population). Participants may have received prior adjuvant chemotherapy/chemoradiation for localized disease if the adjuvant therapy was administered ≥ 6 months prior. All participants must also be naïve to prior endocrine therapy for EC, and confirmed as medically postmenopausal to be eligible.

The study will comprise a Screening Period of up to 28 days in duration; a Study Treatment Phase; a Safety Follow-up Period spanning the time of study treatment discontinuation-including discontinuation due to confirmed disease progression, as applicable-through 28 days after the participant's last dose of any study intervention or the start of subsequent anticancer therapy (whichever occurs first); and a Survival Follow-up Period that will continue until the participant's death or until at least 50% of all study participants have died (whichever occurs first).

While receiving their randomized assigned study treatment, participants will undergo imaging assessments via computed tomography (CT) of the chest/abdomen/pelvis with contrast- or, if CT is medically contraindicated (eg, due to iodine allergy), via magnetic resonance imaging (MRI) with gadolinium-every 8 weeks for the first 12 months and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if they meet all of the following criteria, as applicable:

Applicable to All Participants

1. Is capable of providing signed informed consent as described in Section 10.1.1, which includes compliance with the requirements and restrictions listed in the study informed consent form (ICF) and in this protocol.
2. Is at least 18 years of age, or the legal age of consent in the jurisdiction in which the study is taking place, at the time of providing signed informed consent.
3. Has confirmed Grade 1 or Grade 2 (ie, low-grade histology) endometrioid endometrial adenocarcinoma.

   • Note: Mixed tumor histology is permitted, provided that the non-endometrioid component is < 5%.
4. Is treatment-naïve for Endometrial Cancer (EC) in the advanced/metastatic setting.
5. Is naïve to prior endocrine therapy for EC.
6. Has an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
7. Has adequate organ function, as defined by all of the following:

   * Absolute neutrophil count ≥ 1.5 × 10^9/L
   * Platelets ≥ 100 × 10^9/L
   * Hemoglobin ≥ 8.0 g/dL
   * International Normalized Ratio (INR) ≤ 1.5, unless participant is receiving chronic anti-coagulation therapy as noted below.

   Note: Therapeutic INR is higher in individuals on chronic anti-coagulation treatment. Any such participant whose INR exceeds 1.5 may be considered eligible per Investigator judgment if otherwise meeting the study entry criteria.
   * Creatinine clearance (CLcr) ≥ 45/mL/min, as estimated by Cockcroft-Gault equation
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) both < 2.5 × the upper limit of normal (ULN)
   * Total bilirubin ≤ 1.5 × ULN, in participants with well-documented absence of Gilbert's Syndrome
8. Has QTc interval with Fridericia's correction (QTcF) of < 480 ms
9. Is able to swallow oral medications (or, for selected participants, to receive them by PEG tube as noted below).

   • Note: At the discretion of the Investigator, selected participants with a percutaneous endoscopic gastrostomy (PEG) tube may be eligible. For any such participant, the PEG must allow for the safe and adequate administration of tablets (ie, without crushing or otherwise damaging them).
10. Has a life expectancy of at least 12 weeks.
11. Is medically postmenopausal, as confirmed by the Investigator by meeting one or more of the following criteria:

    * Has undergone bilateral oophorectomy.
    * Is ≥ 60 years of age.
    * Is < 60 years of age and without menses for ≥ 1 year, in the absence of ovarian suppression agents, chemotherapy, tamoxifen, or other agents which may interfere with ovarian function, with laboratory confirmation by Follicle Stimulating Hormone (FSH).
12. If Screening pregnancy testing is clinically indicated per judgment of the Investigator, must have a negative pregnancy test at Screening
13. Must adhere to contraceptive use consistent with local regulations regarding the methods of contraception for those participating in clinical studies
14. Agrees not to donate ova (as applicable) from the time of the first administration of any study intervention until 28 days after the last dose of any study intervention.

    Applicable to Participants with Recurrent Disease
15. Participants with recurrent disease should meet all of the following criteria:

    * Has disease that is measurable according to RECIST v1.1 and outside an irradiated field.
    * Is not eligible for curative intent therapy.
    * Has not received prior anticancer therapy in the recurrent setting.

    Note:

    • Participants are permitted to have received prior adjuvant chemotherapy and/or radiation therapy, provided that such therapy was completed ≥ 6 months before study enrollment

    Applicable to Participants with Advanced/Metastatic Disease
16. Participants with advanced/metastatic disease should meet all of the following criteria:

    * Has disease that is either:
    * FIGO Stage III/IV, measurable according to RECIST v1.1, and outside an irradiated field (as applicable), or
    * FIGO Stage IVB (either measurable or nonmeasurable).
    * Is not eligible for curative intent therapy.
    * Is considered eligible for hormonal therapy.

Exclusion Criteria:

Participants are excluded from this study if they meet any of the following criteria, as applicable:

Applicable to All Participants

1. Tumor histology includes any non-endometrioid component of ≥ 5%.
2. Has EC that meets either of the following criteria:

   * Is amenable to curative intent therapy (ie, surgery, radiation, etc).
   * Was previously treated with systemic therapy (eg, chemotherapy) in the advanced/metastatic setting.
   * Note: Prior adjuvant chemotherapy is allowed, provided that it was completed ≥ 6 months before study enrollment.
3. Has leptomeningeal carcinomatosis or central nervous system (CNS) metastases, unless the participant meets all of the following criteria:

   * Has completed prior therapy for CNS tumor at least 4 weeks before initiating study treatment.
   * Has stable CNS tumor at Screening.
   * Is not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases.
4. Is known to exhibit loss of retinoblastoma protein (Rb) on genetic testing of tumor tissue, if identified per one of the following methods prior to enrollment (note that Rb testing is not an enrollment requirement):

   * PCR
   * Next-generation sequencing
   * Peripheral blood testing
5. Currently has, or has had within the past 3 years, any invasive cancer, except the following:

   * Any prior in situ cancer treated with curative intent
   * Non-melanoma skin cancer, including basal cell carcinoma of the skin
6. Has undergone major surgical intervention within 21 days prior to study entry or minor surgical intervention within 14 days prior to study entry, or is expected to undergo either at any time during the study.
7. Has received within 21 days prior to study entry, is currently receiving, or is expected to receive at any time during the study any radiation therapy, except as palliative therapy for a solitary nontarget lesion.
8. Has received within the 6 months prior to study entry any anti-PD-1/anti-PD-L1 checkpoint inhibitor therapy for any disease.
9. Is currently receiving any of the following substances, and the substance cannot be discontinued within 14 days prior to the first administration of any study intervention:

   * Known strong or moderate CYP3A inducer or strong inhibitor of CYP3A, with the following exception:
   * Note: Participants may receive strong/moderate CYP3A inducers/inhibitors for short periods of time (ie, ritonavir-based treatments for SARS-CoV-2), but the study drug dosing plan during that period of time must be discussed with the Sponsor Medical Monitor.
   * Substances with a narrow therapeutic window that are predominantly metabolized through CYP3A4/5
10. Is currently receiving, is expected to receive at any time during the study, or has discontinued within 14 days prior to study entry any exogenous reproductive hormone therapy (eg, hormone replacement therapy).
11. Has experienced within the 3 months prior to study entry any thromboembolic event or event of intracranial hemorrhage.
12. Has an ejection fraction (EF) of ≤ 45% on any echocardiogram performed within the past 12 months, or has a documented history of congestive heart failure with reduced EF.
13. Has any clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality.
14. Has a history of prolonged QT syndrome or Torsades de Pointes.
15. Has a history of any of the following:

    * Syncope of cardiovascular etiology
    * Ventricular arrhythmia of pathological origin
    * Sudden cardiac arrest
    * Unprovoked venous thromboembolism or known underlying hypercoagulability, with the following additional consideration:
    * Note: Participants with prior deep vein thrombosis may be eligible, provided that they are currently on a stable dose of an anticoagulant and do not pose a bleeding risk in the opinion of the Investigator.
16. Has evidence of active bacterial infection, fungal infection, or viral infection (including SARS-CoV-2 or uncontrolled human immunodeficiency virus [HIV], as noted below) which would preclude safe enrollment in the judgment of the Investigator.

    * Notes:
    * The study SARS-CoV-2 requirements are determined by institutional standards (and local/country regulations, as applicable).
    * At Investigator discretion, any participant who tests positive and/or is symptomatic for SARS-CoV-2 during Screening may either be excluded from the study or delay enrollment until active infection has been excluded per institutional standards.
    * During the study, any SARS-CoV-2 testing is to be performed as clinically indicated for the individual participant. The Investigator must document the results of all tests performed. Any confirmed infection is to be recorded as an AE or, in the event that clinical manifestation warrants such, recorded and handled as an SAE
    * Participants with uncontrolled HIV may be eligible for re-screening after initiating highly active antiretroviral therapy (HAART).
17. Has interstitial pneumonia, or has severe impairment of lung function as defined by either of the following:

    * Vital capacity and diffusing capacity of the lung for carbon monoxide (DLCO) are

      ≤ 50% of the normal predicted values.
    * Oxygen (O2) saturation at rest in ambient environment is ≤ 88%.
18. Has, or shows evidence of, any other active infection, significant medical illness, serious underlying medical condition, abnormal laboratory finding, or psychiatric illness/social situation that might, in the Investigator's judgment, prevent the participant from receiving study treatment or being followed in this study; or which otherwise renders the participant inappropriate for the study as judged by the Investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-18 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Through study completion, an average of 27 months
  PFS is defined as the time from randomization until the date of document disease progression (per RECIST v1.1) or death

SECONDARY OUTCOMES:
Overall Survival (OS) | Through study completion, an average of 27 months
  OS is measured from the date of randomization until death
Progression Free Survival (PFS) by Investigator | Through study completion, an average of 27 months
  PFS based on RECIST v1.1 and assessed by the Investigator Grade 1 or Grade 2 endometrioid EC.
Patient Reported Outcomes/Quality of Life | Through study completion, an average of 27 months
  Defined as the change from baseline
Safety/Tolerability | Through study completion, an average of 27 months
  Defined as the incidence of adverse events, serious adverse events, clinically significant laboratory abnormalities, clinically significant findings on vital signs, ECGs and physical examinations